CLINICAL TRIAL: NCT04927910
Title: Self-applied Acupressure for Arthralgia-fatigue-sleep Disturbance Symptom Cluster in Breast Cancer Survivors Receiving Aromatase Inhibitors
Brief Title: Self-applied Acupressure for Arthralgia-fatigue-sleep Disturbance in Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID 19 outbreak and manpower issues
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The Huazhong University of Science and Technology Union Shenzhen Hospital (Unknown)
Responsible Party: Principal Investigator, Dr CHENG Huilin, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 01
Record Dates: First submitted 2021-03-29; First posted 2021-06-16 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Breast Neoplasms; Cancer Survivor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- True self-acupressure (Experimental): 1) two individual/group acupressure training sessions over 2 weeks and (2) self-acupressure for 6 weeks.
  Interventions: Other: Ture self-acupressure
- Sham self-acupressure (Sham Comparator): Same protocol to the true self-acupressure group but on the sham acupoints
  Interventions: Other: Sham self-acupressure
- Usual care (Other): General advise on managing symptoms provided by healthcare providers
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Ture self-acupressure — 8-week intervention of self-acupressure on acupoints
  Arms: True self-acupressure
Other: Sham self-acupressure — 8-week intervention of self-acupressure on non-acupoints
  Arms: Sham self-acupressure
Other: Usual care — routine care by hospitals
  Arms: Usual care

SUMMARY:
This study aims to evaluate the feasibility, acceptability and preliminary effects of self-applied acupressure on arthralgia-fatigue-sleep disturbance symptom cluster in breast cancer survivors receiving aromatase inhibitors. This is a preliminary randomized controlled trial, with a three-arm trial design including verum self-acupressure, sham self-acupressure, and usual care. Subjects will include 52 breast cancer survivors who are receiving aromatase inhibitors and have experienced a moderate level of joint pain and at least one of the two symptoms including fatigue and sleep disturbance. Subjects who are randomized to either the verum self-acupressure group (group A) or the sham self-acupressure group (group B) will receive up to 8 weeks of the intervention consisting of two components: (1) two individual/group acupressure training sessions over 2 weeks and (2) self-acupressure for 6 weeks. The method and duration of self-acupressure in the sham group will be the same to those in the verum intervention group. The control group will receive usual care. The outcome measures of this study will be related to feasibility, acceptability and preliminary effects of self-acupressure. Individual in-depth interviews will be conducted with selected participants in group A and B to understand their perceptions and perceived effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria

* Female adult aged 18 and older;
* Clinical diagnosis of early-stage (Stage I, II, or IIIa), hormone-receptor-positive breast cancer;
* Completion of surgery, and/or chemotherapy and/or radiotherapy;
* Currently taking the third generation of AIs (anastrozole, letrozole, or exemestane) for at least 1 month;
* Based on their self-reports of moderate symptoms of joint pain and fatigue or sleep disturbance;
* Willing to comply with the intervention protocol, and
* Being able to communicate in Chinese .

Exclusion Criteria:

* Previous receipt of acupuncture and acupressure within the past six months;
* Currently receiving medications (unchanged for 3 month), physical therapy and other complementary and alternative medicines for the treatment of joint pain, fatigue and sleep disturbance;
* Prior joint surgery or fracture during the past six months;
* Mentally incapable of participating in the study (Hong Kong version of Montreal Cognitive Assessment score<22);and
* Inability to perform self-care (Karnofsky Performance Scale score<70).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 21 (Actual)
Dates: Start 2021-06-05 (Actual); Primary Completion 2022-01-29 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
Feasibility measure | Immediately after completion of the intervention (T1)
  Eligibility rate
Feasibility measure | Immediately after completion of the intervention (T1)
  Recruitment rate
Feasibility measure | Immediately after completion of the intervention (T1)
  Attrition rate
Feasibility measure | Immediately after completion of the intervention (T1)
  Time to complete the recruitment
Feasibility measure | Immediately after completion of the intervention (T1)
  Intervention adherence (using a patient-reported diary to document if the patient has completed the intervention daily, experienced any side effects, any other feelings or thoughts )
Acceptability measure | Immediately after completion of the intervention (T1)
  Appropriateness of the intervention components using a self-developed questionnaire (15 close-ended questions mostly on a scale of 1 to 5, higher score indicating higher acceptability and 3 open-ended questions)

SECONDARY OUTCOMES:
Arthralgia | Baseline(T0) and Immediately after completion of the intervention (T1)
  The Brief Pain Inventory- Short Form to assess joint pain related to aromatase inhibitor-induced arthralgia on a scale of 0=no pain, 10=extreme pain
Fatigue | Baseline(T0) and Immediately after completion of the intervention (T1)
  The Brief Fatigue Inventory to measure fatigue on a scale of 0=no fatigue, 10=extreme fatigue
Sleep disturbance | Baseline(T0) and Immediately after completion of the intervention (T1)
  The Pittsburgh Sleep Quality Index (PSQI) to measure sleep disturbance (with different item options) [a global score ranges from 0 to 21, with a higher score indicating poor sleep quality]
Health-related quality of life | Baseline(T0) and Immediately after completion of the intervention (T1)
  The Functional Assessment of Cancer Therapy scale (FACT-G) to measure health-related quality of life on a scale of 0=lower health-related quality of life, 4=higher health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Huilin Cheng, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Huazhong University of Science and Technology Union Shenzhen Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No